CLINICAL TRIAL: NCT03443362
Title: Prospective, Observational, Longitudinal Cohort Study on the Role of Endothelial Cells in the Pathogenesis of Chronic Urticaria.
Brief Title: Role of Endothelial Cells in the Pathogenesis of Chronic Urticaria.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Olivier Michel (Other)
Responsible Party: Sponsor-Investigator, Olivier Michel, Head of clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-Chronic urticaria
Record Dates: First submitted 2018-02-16; First posted 2018-02-23 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Chronic Urticaria
Keywords: Chronic Urticaria; Endothelial cells
MeSH Terms: conditions — Chronic Urticaria | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skin specimens (3 mm punch biopsy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic urticaria: 50 consecutive chronic urticaria patients receiving medical care within the CHU Brugmann Hospital. Diagnose according to the European Academy of Allergy and Clinical Immunology (EAACI) guidelines.
  Interventions: Procedure: Punch Biopsy; Procedure: Blood sampling
- Control: 20 healthy control patients, without chronic urticaria. Patients coming to the CHU Brugmann hospital for the excision of atypical naevi.
  Interventions: Procedure: Punch Biopsy; Procedure: Blood sampling

INTERVENTIONS:
Procedure: Punch Biopsy — A 3 mm punch biopsy will be taken from lesional and non-lesional skin as a routine procedure.
Procedure: Blood sampling — Blood sampling

SUMMARY:
Chronic urticaria (CU) is a disease that usually affects a large visible amount of surface of the skin. It is accompanied by severe itch and feeling of burned skin. Therefore the disease has a big impact on the quality of life of patients. Unfortunately, to date CU is not easily controlled by its few existing treatment options (i.e. antihistamines, omalizumab, cyclosporine).

This research's main perspective is to improve quality of life for CU patients by first of all focusing on a good clinical diagnosis of (different subtypes of) CU in a CU reference center, and secondly by gaining more insight on the pathogenesis of the disease to expand knowledge on potential new targeted treatments for the patients.

DETAILED DESCRIPTION:
Chronic urticaria (CU) is an inflammatory skin disease that is defined by the presence of urticaria (hives), on most days of the week, for a period of six weeks or longer. About 40 percent of patients with CU have accompanying episodes of angioedema. It is classified as chronic inducible urticaria (CIU) in which urticaria is induced by one or more environmental stimuli (such as heat, cold, pressure applied to the skin, exercise, water, vibration, and sunlight) and chronic spontaneous urticaria (CSU) which refers to CU in which appearance of lesions is not triggered by consistent or identifiable factors. At any given time, CU affects up to 1 percent of the general population in the United States, and the prevalence is believed to be similar in other countries. So far, epidemiological studies for a Belgian population haven't been performed yet.

It is generally proposed that patients with CU have defects in mast cell and/or basophil trafficking, signaling and/or function. Nevertheless more recently also other cells seem to be involved: lymphocytes, eosinophils, endothelial cells (ECs). The integrity of EC structure and function is important in the maintenance of the vessel wall and circulatory function. As a barrier, the endothelium is semi-permeable and controls molecular transport between the blood and the tissues. Under basal conditions, ECs are involved in maintaining the anti-thrombotic blood-tissue interface by regulating thrombosis, thrombolysis, platelet adherence, vascular tone and blood flow. In CU, mast cells are activated and histamine release occurs. This histamine binds to its receptor on the ECs causing vasodilation and extravasation. This endothelial function/dysfunction can be characterized by several biological markers from different signalization/activation pathways. Vascular injury induces release of vascular endothelial growth factor (VEGF) to stimulate angiogenesis. Cytokine stimulation triggers the expression and release of adhesion molecules (e.g., E-selectin, ICAM-1, VCAM-1), making transendothelial migration of lymphocytes possible. In particular, E-selectin is expressed only by activated endothelium; however, its circulating form (sE-selectin) can be found in the plasma after enzymatic cleavage or from shedding by damaged or active ECs. Furthermore it is known for ECs to interact with mast cells through the production of Stem Cell Factor (SCF; c-kit ligand) to influence mast cell proliferation and differentiation. Asero et al (2003) determined serum SCF levels in 65 CIU patients and found no difference from those found in healthy controls. Nevertheless, the increase in mast cells in skin biopsy specimens, along with the absence of systemic eosinophilia in CIU patients suggests a possible role for stem cell factor (SCF) in CU pathogenesis.

Endothelial progenitor cells (EPC) normally have the ability to develop into fully mature EC and contribute to neovascularization by targeting sites of endothelial injury. Furthermore it is shown that acute exercise-induced nitric oxide production contributes to upregulation of circulating endothelial progenitor cells in healthy subjects. Since exercise is a known trigger for CU, it would be interesting to investigate the effect of exercise on EPC recruitment and EC activation in CSU.

Microvascular damage and EC injury is described in multiple diseases such as diabetes and scleroderma. This can be evaluated by nail fold videocapillaroscopy (NVC). The integrity of vessel walls is compromised in CU, of which the appearance of wheals due to the extravasation process seems to be the most obvious symptom clinically. It would be interesting to examine if there are microscopical abnormalities on NVC that could help identify (certain subtypes of) CU. If present, correlations between these abnormalities and disease severity can be further investigated.

The objectives of the study are:

* To determine the incidence of CU (CSU and CIU) in a Belgian city center hospital
* To investigate the role of ECs in CSU on a clinical and molecular level

ELIGIBILITY:
Inclusion Criteria:

All patients diagnosed with chronic urticaria receiving medical care within the CHU Brugmann Hospital. Diagnose performed according to the European Academy of Allergy and Clinical Immunology (EAACI) guidelines.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a diagnose of chronic urticaria receiving medical care within the CHU Brugmann Hospital. Diagnose performed according to the European Academy of Allergy and Clinical Immunology (EAACI) guidelines.
  The control group consists in patients beeing followed within the CHU Brugmann Hospital for the ellipsoid excision of atypical naevi on remnant healthy skin.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Stem cell factor expression | 6 months
  Immunohistochemistry performed on cryostat sections with a monoclonal antibody
E-selectin expression | 6 months
  Immunohistochemistry performed on paraformaldehyde fixed sections with a monoclonal antibody
Vascular endothelial growth factor (VEGF) expression | 6 months
  Immunohistochemistry performed with a monoclonal antibody on paraffin sections
C5B9 complement complex expression | 6 months
  Immunofluorescence staining performed on paraffin-embedded tissue blocks

SECONDARY OUTCOMES:
Incidence of chronic inducible urticaria | 6 months
  Incidence of chronic inducible urticaria within the CHU Brugmann Hospital. Diagnose established by means of provocation tests.
Incidence of chronic spontaneous urticaria | 6 months
  Incidence of chronic spontaneous urticaria within the CHU Brugmann Hospital. Diagnose established by means of provocation tests.

CONTACTS AND LOCATIONS:
Overall Officials: Yora Mostmans, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaplan AP. Chronic urticaria: pathogenesis and treatment. J Allergy Clin Immunol. 2004 Sep;114(3):465-74; quiz 475. doi: 10.1016/j.jaci.2004.02.049. PMID 15356542
- [Background] Zuberbier T, Aberer W, Asero R, Bindslev-Jensen C, Brzoza Z, Canonica GW, Church MK, Ensina LF, Gimenez-Arnau A, Godse K, Goncalo M, Grattan C, Hebert J, Hide M, Kaplan A, Kapp A, Abdul Latiff AH, Mathelier-Fusade P, Metz M, Saini SS, Sanchez-Borges M, Schmid-Grendelmeier P, Simons FE, Staubach P, Sussman G, Toubi E, Vena GA, Wedi B, Zhu XJ, Nast A, Maurer M; Dermatology Section of the European Academy of Allergy and Clinical Immunology; Golbal Allergy and Asthma European Network; European Dermatology Forum; World Allergy Organization. Methods report on the development of the 2013 revision and update of the EAACI/GA2 LEN/EDF/WAO guideline for the definition, classification, diagnosis, and management of urticaria. Allergy. 2014 Jul;69(7):e1-29. doi: 10.1111/all.12370. PMID 24898678
- [Background] Greaves M. Chronic urticaria. J Allergy Clin Immunol. 2000 Apr;105(4):664-72. doi: 10.1067/mai.2000.105706. PMID 10756214
- [Background] Gaig P, Olona M, Munoz Lejarazu D, Caballero MT, Dominguez FJ, Echechipia S, Garcia Abujeta JL, Gonzalo MA, Lleonart R, Martinez Cocera C, Rodriguez A, Ferrer M. Epidemiology of urticaria in Spain. J Investig Allergol Clin Immunol. 2004;14(3):214-20. PMID 15552715
- [Background] Hellgren L. The prevalence of urticaria in the total population. Acta Allergol. 1972;27(3):236-40. doi: 10.1111/j.1398-9995.1972.tb01420.x. No abstract available. PMID 4678809
- [Background] Zuberbier T, Balke M, Worm M, Edenharter G, Maurer M. Epidemiology of urticaria: a representative cross-sectional population survey. Clin Exp Dermatol. 2010 Dec;35(8):869-73. doi: 10.1111/j.1365-2230.2010.03840.x. PMID 20456386
- [Background] Sumpio BE, Riley JT, Dardik A. Cells in focus: endothelial cell. Int J Biochem Cell Biol. 2002 Dec;34(12):1508-12. doi: 10.1016/s1357-2725(02)00075-4. PMID 12379270
- [Background] Constans J, Conri C. Circulating markers of endothelial function in cardiovascular disease. Clin Chim Acta. 2006 Jun;368(1-2):33-47. doi: 10.1016/j.cca.2005.12.030. Epub 2006 Mar 10. PMID 16530177
- [Background] Coleman JW, Holliday MR, Kimber I, Zsebo KM, Galli SJ. Regulation of mouse peritoneal mast cell secretory function by stem cell factor, IL-3 or IL-4. J Immunol. 1993 Jan 15;150(2):556-62. PMID 7678275
- [Background] Asero R, Tedeschi A, Lorini M, Gerosa M, Meroni P, Riboldi P. Circulating stem cell factor in patients with chronic idiopathic urticaria. Ann Allergy Asthma Immunol. 2003 Jul;91(1):79-81. doi: 10.1016/S1081-1206(10)62063-7. PMID 12877454
- [Background] Kuwana M, Okazaki Y. Quantification of circulating endothelial progenitor cells in systemic sclerosis: a direct comparison of protocols. Ann Rheum Dis. 2012 Apr;71(4):617-20. doi: 10.1136/annrheumdis-2011-200713. Epub 2012 Jan 17. PMID 22258488
- [Background] Yang Z, Wang JM, Chen L, Luo CF, Tang AL, Tao J. Acute exercise-induced nitric oxide production contributes to upregulation of circulating endothelial progenitor cells in healthy subjects. J Hum Hypertens. 2007 Jun;21(6):452-60. doi: 10.1038/sj.jhh.1002171. Epub 2007 Mar 15. PMID 17344910
- [Background] Fletcher GF, Balady GJ, Amsterdam EA, Chaitman B, Eckel R, Fleg J, Froelicher VF, Leon AS, Pina IL, Rodney R, Simons-Morton DA, Williams MA, Bazzarre T. Exercise standards for testing and training: a statement for healthcare professionals from the American Heart Association. Circulation. 2001 Oct 2;104(14):1694-740. doi: 10.1161/hc3901.095960. No abstract available. PMID 11581152
- [Background] Cutolo M, Sulli A, Pizzorni C, Smith V. Capillaroscopy as an Outcome Measure for Clinical Trials on the Peripheral Vasculopathy in SSc-Is It Useful? Int J Rheumatol. 2010;2010:784947. doi: 10.1155/2010/784947. Epub 2010 Aug 16. PMID 20827384
- [Derived] Mostmans Y, De Smedt K, Feoli F, Waelput W, De Maertelaer V, Olemans C, Meiers I, Cielen T, Corazza F, Michel O, Richert B. Elevated cutaneous expression of stem cell factor in chronic spontaneous urticaria: a prospective cohort study. Clin Exp Dermatol. 2024 Nov 22;49(12):1659-1667. doi: 10.1093/ced/llae252. PMID 38963799